CLINICAL TRIAL: NCT06590727
Title: Resources Assessment to Increase pSychological dEvelopment in Breast Cancer Patients
Brief Title: Psychological Well-being in Patients With Breast Cancer
Acronym: RAISE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6470
Record Dates: First submitted 2024-05-24; First posted 2024-09-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Distress Thermometer — Enrolled patients will be given a clinical psychological interview. Then they will be given an anamnestic interview and the aforementioned questionnaires will be administered.
  Other Names: Hospital Anxiety and Depression Scale; Mini Mental of Adjustment for Cancer Scale; Clinical Outcomes in Routine Assessment; Post-traumatic growth inventory

SUMMARY:
Psychoncological evaluation in patients diagnosed with breast cancer is often limited to psychological distress and does not include evaluation of individual resources. This assessment could contribute to implement adherence to treatment protocols and eventual post traumatic growth. This study shows a new model of psychoncological triage by screening the risk of psychological distress and coping resources in patients with non metastatic breast cancer while waiting for surgery. The evaluation is performed at the hospital after the diagnosis and by means of psychological counseling and psychodiagnostic assessment (T0) with follow up interventions along the continuum of care.

Recruitment of the sample will take place in three different phases. It Includes time zero (T0) when patients are assessed during the pre-hospitalisation pathway. Time 1 (T1) patients are re-evaluated during the perioperative hospitalisation phase. Time 2 (T2) patients are re-evaluated after nine months at the end of treatment. As this phase is highly individualised for each patient and therefore susceptible to variation in duration and treatment modalities. Online psychometric revaluation will be possible. The link to the questionnaires will be sent to patients by e-mail and subsequently by telephone or in person contact.

Patients are evaluated by following questionnaires. Distress Thermometer (DT). Hospital Anxiety and Depression Scale (HADS). Mini Mental of Adjustment for Cancer Scale (MINIMac) and Clinical Outcomes in Routine Assessment (CORE OM) and Post Traumatic Growth Inventory

Cut off COREOM is From 10 to 15 Mild. From 15 to 20 Moderate. From 20 to 25 Mod or Severe. From 25 Severe. Scoring is from 0 is not at all and to 4 is very often/always. Reversed items 3.4. 7. 12. 19. 21. 31. 32. Higher scores correspond to greater problems.

The cut off of the distress thermometer is greater than 4. The cut off oh HADS is 7. From 0 to 7 is considered normal. A score of 8 or higher indicating probable presence of a mood disorder.

The miniMAC scale is a self-descriptive tool. The respondent on his or her own evaluates, using a four point scale to what extent a given statement applies to him or her at present. Each statement is rated on a scale of 1 (definitely not) to 4 (definitely yes), and the results available for each of the four strategies for dealing with the disease are 7-28 points. The higher the score, the greater the severity of the behaviors in the patient's struggle with cancer.

Post Traumatic Growth Inventory. Each of the 21 items falls under one of the five factors and are scored accordingly. A summation of the scores indicates the level of post-traumatic growth.

The advantage of this scale is that the categorization of scores according to the five factors are suggestive of which area of self-development is predominant in us and which area might be a little behind.

ELIGIBILITY:
Inclusion Criteria:

* 18 years
* candidates for surgery
* candidates for adjuvant and/or neoadjuvant treatment

Exclusion Criteria:

* 0 to 17 years old
* severe language deficits
* severe barriers
* Patients unable to understand and express informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who have been diagnosed with breast cancer. They will be considered in a retrospectively patients who have already accessed (2022-2023) and prospectively those who will access in the future (2024-2026) the services of:
  UOC Senologic Surgery, UOS Integrated Therapies in Senology, UOS of Clinical Psychology FPG IRCSS to perform routine screening, psychometric evaluation, or psychological intake.
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Patients assessment | 1 year
  Evaluate the information coming from the multidimensional evaluation (for example clinical or laboratory and psychometric evaluations) of the cancer patient during his diagnostic and therapeutic process at the Fondazione Policlinico Universitario Agostino Gemelli IRCCS.

SECONDARY OUTCOMES:
Psychological distress | 1 year
  Investigate the risk of psychological distress of the cancer patient through the results reported in the study questionnaires
Factors predictive | 1 year
  Quickly identify the predisposition to states of anxiety and depression through the detection of predictive factors that emerged from the evaluation of the study questionnaires administered to the cancer patient.
Coping strategies | 1 year
  Evaluate the presence of coping strategies that the cancer patient is able to implement during the treatment process by reading the study questionnaires administered three times
Identifying possible correlations | 1 year
  Identifying possible correlations between personological, emotional and behavioural characteristics, coping styles and possible anxious-depressive symptoms and psychological distress psychological distress;
Personalised care pathway | 1 year
  Identify a personalized care path for the cancer patient followed in the study, based on the evaluation of the overall results of the questionnaires administered and the overall psychological evaluation that emerged.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Belella, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOS Psicologia Clinica, Roma, Italy